CLINICAL TRIAL: NCT03726216
Title: Observational Study on the Use of Xydalba: A Multicenter, Prospective Study to Characterize the Use of Xydalba in France
Brief Title: Xydalba Utilization Registry in France
Status: Completed | Type: Observational
Sponsor: Correvio International Sarl (Industry)
Collaborators: Universal Medical Group (Unknown); PrimeVigilance (Industry)
Responsible Party: Sponsor
Organization: Advanz Pharma (Industry)
Other Study IDs: DAL-REG01-FRA
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2020-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — dalbavancin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- use of Xydalba, >18 years: Male and female patients, ≥18 years of age at the time of receipt of Xydalba. Patients who received at least one Xydalba administration in France
  Interventions: Drug: Xydalba

INTERVENTIONS:
Drug: Xydalba — Information will be recorded about Xydalba administration (e.g. dose(s), number of infusions, length of infusions, dates or schedule of administration, sites of administration [e.g. hospital, ICU]), and reason for discontinuation, including response to treatment to assess whether the patient was clinically improving when Xydalba was discontinued
  Other Names: Dalbavancine

SUMMARY:
This observational study will collect data on the use of the drug Xydalba® in daily clinical practice in France. Such observational studies are also referred to as registries. The sponsor of the study is Correvio International Sárl, based in Switzerland.

Xydalba® contains the active substance dalbavancin, a remedy for a certain type of bacterial pathogens (so-called "gram positive bacteria") which cause the disease. Active ingredients against bacteria are also called antibiotics.

Correvio wants to know which patients received the drug and how the disease went. The treatment places where you got Xydalba, ie clinic, intensive care unit or elsewhere should be recorded. In addition, it is important in this type of medication to track whether the pathogens are changing in any way. Any safety-relevant events (such as side effects) that have occurred during treatment should be investigated by the sponsor and submitted to the competent European authorities.

DETAILED DESCRIPTION:
OBJECTIVES

The objectives of this registry are as follows:

* To determine the following characteristics in patients who received intravenous Xydalba administration:
* Patient characteristics.
* Disease characteristics.
* Pathogen characteristics.
* To characterize the usage of Xydalba.
* To characterize the patient's residence and, in hospitalized patients, the lengths of hospital and intensive care unit (ICU) stays, and the destination upon hospital discharge.
* To assess the response of Xydalba treatment, based on clinician determination.
* To characterize the major healthcare resource utilization (HRU) of patients treated with Xydalba.

REGISTRY DESIGN:

This is a multicenter, prospective registry of adult patients treated with Xydalba in France.

All Adverse events (AEs) (serious and non-serious; special situations; related and not-related, collected prospectively or retrospectively) will be recorded in the eCRF. Treatment related AEs and SAEs will be reported to the healthcare authorities, as requested by local regulations and according to current Guideline on good pharmacovigilance practices (GVP) Module VI - Collection, management and submission of reports of suspected adverse reactions to medicinal products (Rev 2).

TEST PRODUCT (S), DOSE, AND MODE OF ADMINISTRATION Xydalba (dalbavancin) as prescribed by the physician according to clinical practice.

RATIONALE:

This prospective registry is designed to capture information about the clinical use of Xydalba, its safety and effectiveness, characteristics of the patient, disease, pathogen, clinical course, treatment course, and hospitalization. This registry will capture the data in real world setting on patients who received Xydalba.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient associate to a social protection scheme, ≥18 years of age at the time of receipt of Xydalba
* The patient received at least one infusion of Xydalba
* Patient signed the consent form

Exclusion Criteria:

* The patient was enrolled in a clinical trial in which treatment for Xydalba is managed through a protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The registry will capture the data in real world setting on patients who received at least one does of Xydalba.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Clinical response | 30 days
  Prevalence of ABSSSI and other primary diagnoses among patients who received Xydalba (dalbavancin) as treatment for this primary diagnosis

SECONDARY OUTCOMES:
Clinical response by diagnosis | 30 days
  Clinical response by cured, improved, failure, non-evaluable, worsening or other (non-clinically evaluable)
Clinical response by diagnosis | 30 days
  Clinical response by diagnosis (ABSSSI, Gram-positive bacteremia, other associated diagnosis)
Time from Xydalba treatment onset to clinical response | 30 days
Adverse Events, Adverse Drug Reactions and Special Situations | 30 days

OTHER OUTCOMES:
Xydalba Treatment dose(s) | 30 days
  Dose(s) of Xydalba in mg per infusion
Number of Xydalba Infusions | 30 days
  number of Infusions given
Length of Xydalba Infusions | 30 days
  length of Infusions in minutes
Days of Xydalba treatment | 30 days
  number of Days of treatment
Percentage of monotherapy vs. concurrent therapy | 30 days
  % of cases for which Xydalba is given as monotherapy and % of cases for which Xydalba is given as concurrent therapy
Percentage first-line vs. subsequent-line monotherapy | 30 days
  % of cases for which Xydalba is given as first-line and % of cases for which Xydalba is given as subsequent-line
Prior Antibiotic Therapies | 30 days
  Descriptive summary of other antibiotic therapies received
Reason for discontinuation | 30 days
  descriptive listing of type of reasons

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Centre hospitalier d'Ajaccio, Maladies infectieuses et tropicales, Ajaccio
  - Centre Hospitalier Universitaire de Bordeaux, Hopital Saint-André, Bordeaux
  - CHU Bordeaux Pellegrin, Bordeaux
  - Hôpital Raymond-Poincaré, Garches
  - CHU GRENOBLE, Maladies infectieuses et tropicales, Grenoble
  - Hôpital de la Croix-Rousse, Service des maladies infectieuses et tropicales, Lyon
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Centre hospitalier régional et universitaire de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Centre hospitalier universitaire de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes (CHU), Nîmes
  - Hôpital Ambroise-Paré,Maladies infectieuses, Paris
  - Pontchaillou University Hospital, Infectious Diseases and Intensive Care Unit, Rennes
  - Centre hospitalier universitaire de Saint-Étienne, Saint-Etienne
  - Centre Hospitalier de Tourcoing,Service des Maladies Infectieuses et du Voyageur, Tourcoing

IPD SHARING:
Plan to Share IPD: No